CLINICAL TRIAL: NCT03060291
Title: Prevention of Substance Use in At-Risk Students: A Family-Centered Web Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Beth Stormshak, Knight Chair and Professor, College of Education, and Director, Prevention Science Institute, University of Oregon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA037628 (NIH); R01DA037628 (NIH)
Record Dates: First submitted 2017-02-12; First posted 2017-02-23 (Actual); Results first posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-11

CONDITIONS: Substance Use; Conduct Disorders in Adolescence; Depression; Anxiety
Keywords: Family Check-up
MeSH Terms: conditions — Substance-Related Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three conditions: a web/mobile-only condition, a web/mobile + coach condition, or a wait list control group who will receive the web/mobile-only treatment one year after enrolling in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Web/ Mobile-only (Experimental): Participants will complete the FCU online independently, without the help of a coach.
  Interventions: Behavioral: FCU-Online, web/ mobile only
- Web/mobile + coach (Active Comparator): Participants will complete the FCU online and will be contacted by a family coach. The coach will conduct motivational interviewing and provide support to parents via phone. Participants in this condition will have contact with a coach at least 2 times.
  Interventions: Behavioral: FCU-Online, web/ mobile + coach
- Wait list control (No Intervention): Participants in this condition will receive "middle school as usual", meaning that they will continue to receive whatever services are normally provided by the middle school during the year of their participation in the study. Once their research participation is completed (i.e., after they complete their final follow-up survey), participants in this condition will be offered the opportunity to use the FCU-Online website if they wish, without the support of a coach. No additional data will be collected.

INTERVENTIONS:
Behavioral: FCU-Online, web/ mobile only — Participants will be invited to complete the FCU via the FCU-Online website. They will complete an assessment, receive computer-generated feedback, and access to skills units designed to teach parents the importance of using specific parenting skills, provide practice opportunities to try these skills, and tools to track their use of these parenting skills and any associated changes in child behavior.
  Arms: Web/ Mobile-only
Behavioral: FCU-Online, web/ mobile + coach — Participants will be invited to complete the FCU via the FCU-Online website. They will complete an assessment, receive computer-generated feedback, and access to skills units designed to teach parents the importance of using specific parenting skills, provide practice opportunities to try these skills, and tools to track their use of these parenting skills and any associated changes in child behavior. Participants will also have access to a "family coach" who will motivate parents to enhance parenting skills and provide support while they are learning to use these skills.
  Arms: Web/mobile + coach

SUMMARY:
The purpose of this study is to develop and evaluate the effectiveness of a web-based version of the Family Check-up (FCU). The FCU is a school-based family-centered intervention that has been developed over the past 20 years and tested across the United States with diverse populations. It focuses on enhancing parenting skills and family management in early adolescence. The FCU has been shown to be highly effective at reducing adolescent problem behavior, achievement problems, depression, and substance use over an extended period of time.

In the original FCU, parents complete an assessment that evaluates family strengths and challenges. They then receive feedback from a family consultant about how their data compare to other families with children of the same age. As part of this feedback session, the consultant helps motivate parents to make changes at home that will positively impact their child and family overall. Parents and consultants decide together which child behaviors they most want to see change. The consultant then works with parents to enhance relevant parenting and family management skills.

Despite the demonstrated effectiveness of this intervention, few schools have the resources and staffing to implement it without substantial support. It seems, then, that schools would benefit from an online package that requires fewer school resources to implement. The FCU-Online is designed to incorporate the successful components of the original FCU while reducing the burden on schools. And, because it is accessed online, parents can utilize this resource at a time and location convenient to them.

In this study, 300 families will be randomly assigned to one of three conditions: a web/ mobile-only version of the FCU, a web/mobile + coach version, or middle school as usual. Research on mental health interventions delivered over the internet suggests that a coach or "in-person" contact enhances outcomes. However, programs that require no coaching or in-person contact are cheaper and easier for schools to deliver. Therefore, a web/ mobile-only version may allow more schools to deliver the intervention to a greater number of families and children. Thus, investigators will test the relative effectiveness of a coach version versus an online-only version at improving key parenting skills. It is predicted that changes in parenting will lead to reductions in risk behavior, such as problem behavior at school and substance use.

DETAILED DESCRIPTION:
School-based, family-centered interventions for reducing substance use in adolescence have been shown to be highly effective and result in reductions in problem behavior, achievement problems, depression, and substance use over time. Although these interventions have been shown to be effective in efficacy trials across the United States, few schools have the resources to implement these interventions without substantial support. Barriers such as low staffing, poorly trained staff, and limited resources prevent the successful uptake of family-centered interventions in schools, yet most school systems are supportive of enhancing family-school partnerships. Because school systems lack the necessary infrastructure and resources to deliver such an intervention, they would benefit from an online package that is evidence based and accessible to parents. However, few family-centered, web-based interventions for substance use prevention exist on the Internet, and few if any are derived from empirically based programs.

To address this gap, project investigators are developing and will be testing the efficacy of an online version of the Family Check-Up (FCU) for schools that parents can use either at the school or at home. The FCU is a school-based, model-driven intervention that has been developed during the past 20 years and has been iteratively revised on the basis of multiple intervention trials with diverse populations. This study is building upon the investigators' successful program of research by developing and testing the efficacy of The FCU-Online. It is designed to incorporate the successful components of the original FCU, such as a strengths-based assessment that is norm referenced, feedback using motivational interviewing, and follow-up modules that focus on enhancing parenting skills and family management in early adolescence. This research is designed to randomly assign 300 families to receive middle school as usual, the FCU-Online web/mobile only, or the FCU-Online web/mobile+coach version. Research on the delivery of mental health interventions via the Internet suggests that a coach or "in person" contact enhances outcomes; however, programs that require no coaching or in-person contact may have a larger public health impact. A coach version of the intervention will be compared with an online-only version that requires no staffing at schools. Project investigators will test the efficacy of this online version with respect to changing key parenting constructs, such as positive parenting and parental monitoring. It is predicted that changes in parenting will lead to reductions in risk behavior, such as problem behavior at school and substance use. This research will significantly contribute to researchers' understanding of effective interventions for adolescents that reduce risk behavior and substance use during the transition to high school, and it can significantly contribute to the overall uptake and dissemination of family-centered interventions in schools.

Specific aims of this study are as follows:

Aim 1: Design and evaluate a web-based FCU intervention for at-risk families of early adolescents (ages 11-14) that is guided by feedback from focus groups and targets known risk factors of later substance use. The program will feature online assessment and feedback to caretakers delivered via either phone or Internet. An intervention website application and mobile messaging will support delivery of program modules and help motivate and facilitate tracking of activities. Examples will be presented to potential users, including parents and school personnel, to assess feasibility and usability. A 6-month pilot study will test all recruitment, assessment, and intervention procedures.

Aim 2: Examine the efficacy of the FCU-Online intervention by conducting a randomized, controlled trial of 300 at-risk middle school youths. Research suggests that a live coach enhances outcomes associated with web-based interventions; however, a web-based intervention that requires no coaching can be widely disseminated and has greater potential for a large public health impact. The investigators propose to examine outcomes associated with a web/mobile+coach version and a web/mobile-only version of the FCU. Families will be randomly assigned to the FCU-Online intervention (100 web/mobile+coach, 100 web/mobile only) or middle school as usual (n = 100).

Aim 2.1. Evaluate main effects of both versions of the FCU-Online, including academic achievement, behavioral control, family cohesiveness, and delayed onset of substance use.

Aim 2.2. Test a developmental, mediational model in which parenting skills and behavior mediate changes in youth behavior over time. It is expected that families who receive the FCU will show reductions in growth of youths' risk behavior, compared with the control group. Reductions will be mediated by positive changes in parenting behaviors and parenting skill development.

Aim 2.3. Examine moderators, including gender, ethnicity, and socioeconomic status, and model intervention effects by testing moderators over time. The investigators will assess the feasibility of the FCU as an Internet-delivered intervention in middle schools, the extent to which participants engage in the intervention and complete the program, satisfaction with the program, and effects of the FCU on improved parenting skills, positive youth adjustment, and reductions in youth problem behavior over 2 years.

Aim 2.4. Examine factors related to successful uptake and implementation of the intervention in schools. The public health impact of an Internet intervention is diminished if uptake of the intervention is poor. To understand factors related to implementation in schools, school personnel will be trained at the end of the project in delivery of the FCU-Online intervention. The investigators will assess feasibility, usage, coach fidelity, and uptake through engagement data collected via the website. Data from teachers and school administrators will be collected to examine factors that promote implementation in schools and that further researchers' understanding of how this intervention will be applied in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* enrollment of child in 6th or 7th grade at one of the 6 participating middle schools;
* caregivers are the parent or legal guardian of the participating youth;
* caregivers have web access at home or are willing to access the web via computers located in the school or public library

Exclusion Criteria:

* children with severe developmental disabilities or physical disabilities (e.g., autism, genetic disorders, Down syndrome) will not be eligible to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Stormshak, PhD, Principal Investigator — University of Oregon; John Seeley, PhD, Principal Investigator — University of Oregon
Locations (1):
- University of Oregon, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stormshak E, Connell A, Mauricio AM, McLaughlin M, Caruthers A. Digital Health Delivery of Parenting Skills to Improve Conduct Problems in Middle School Youth Across Two Distinct Randomized Trials. Prev Sci. 2025 May;26(4):582-591. doi: 10.1007/s11121-024-01750-2. Epub 2024 Nov 18. PMID 39556238
- [Derived] Danaher BG, Seeley JR, Stormshak EA, Tyler MS, Caruthers AS, Moore KJ, Cardenas L. The Family Check-Up Online Program for Parents of Middle School Students: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Jul 18;7(7):e11106. doi: 10.2196/11106. PMID 30021712

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During two consecutive school years, all families with a 6th or 7th grade student enrolled in one of eight public middle schools in Oregon (two rural, two urban, and four suburban schools) were contacted and invited to participate via an email sent by the principal. Schools ranged in size from 294 to 839 students; the percentage of students qualifying for free or reduced lunch ranged from 52% to 100%. Families were recruited between February 2017 and June 2018.
Pre-assignment Details: 432 families inquired about study participation. Some were excluded due to not returning the initial survey (n=66), declining to participate (n=8), or not meeting inclusion criteria (n=11). Siblings, monolingual Spanish speakers, and families who participated in prior FCU studies (n=25) were assigned to a nonexperimental condition; they received support but were not included in the analytic sample. Families who returned baseline surveys (n=322) were randomly assigned to one of three conditions.
Period: Baseline
Arm/Group | Web/ Mobile-only | Web/Mobile + Coach | Wait List Control
Started | 109 | 108 | 105
Completed | 109 | 108 | 105
Not Completed | 0 | 0 | 0
Period: 3-month Follow-up
Arm/Group | Web/ Mobile-only | Web/Mobile + Coach | Wait List Control
Started | 109 | 108 | 105
Completed | 101 | 98 | 103
Not Completed | 8 | 10 | 2
Not completed — Declined to respond | 8 | 10 | 2
Period: 6-month Follow-up
Arm/Group | Web/ Mobile-only | Web/Mobile + Coach | Wait List Control
Started | 109 | 108 | 105
Completed (Because no families were ever lost to follow-up or withdrew from the study, all families who participated at baseline were invited to participate at each follow-up wave. Thus, there are a a few families who participated at 6-month or 12-month follow-up who did not participate at an earlier follow-up wave.) | 102 | 95 | 101
Not Completed | 7 | 13 | 4
Not completed — Declined to respond | 7 | 13 | 4
Period: 12-month Follow-up
Arm/Group | Web/ Mobile-only | Web/Mobile + Coach | Wait List Control
Started | 109 | 108 | 105
Completed (Because no families were ever lost to follow-up or withdrew from the study, all families who participated at baseline were invited to participate at each follow-up wave. Thus, there are a a few families who participated at 6-month or 12-month follow-up who did not participate at an earlier follow-up wave.) | 102 | 92 | 99
Not Completed | 7 | 16 | 6
Not completed — Declined to respond | 7 | 16 | 6

BASELINE CHARACTERISTICS:
Population: At baseline there were 109 parent-child dyads in the web/ mobile-only condition (n=218), 108 dyads in the web/ mobile + coach condition (n=216), and 105 dyads in the wait list control condition (n=210). Descriptive statistics have been provided for the children's demographics, but only parent data were included in outcome analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Web/ Mobile-only | Web/Mobile + Coach | Wait List Control | Total
Number analyzed (Participants) | 218 | 216 | 210 | 644
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: At baseline there were 109 parent-child dyads in the web/ mobile-only condition, 108 dyads in the web/ mobile + coach condition, and 105 dyads in the wait list control condition. Data entered in this section represent individuals, not dyads. Child demographics were collected but only parent outcomes analyzed.
  years
    parent: number analyzed (Participants) | 109 | 108 | 105 | 322
    parent | 40.27 (6.18) | 40.11 (6.24) | 40.23 (6.32) | 40.20 (6.23)
    child: number analyzed (Participants) | 109 | 108 | 105 | 322
    child | 11.83 (0.69) | 11.87 (0.76) | 11.93 (0.68) | 11.88 (0.71)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: At baseline there were 109 parent-child dyads in the web/ mobile-only condition, 108 dyads in the web/ mobile + coach condition, and 105 dyads in the wait list control condition. Data entered in this section represent individuals, not dyads. Child demographics were collected but only parent outcomes analyzed.
  Participants
    parent: number analyzed (Participants) | 109 | 108 | 105 | 322
    parent: Female | 93 | 102 | 96 | 291
    parent: Male | 16 | 6 | 9 | 31
    child: number analyzed (Participants) | 109 | 108 | 105 | 322
    child: Female | 54 | 51 | 49 | 154
    child: Male | 55 | 57 | 56 | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: At baseline there were 109 parent-child dyads in the web/ mobile-only condition, 108 dyads in the web/ mobile + coach condition, and 105 dyads in the wait list control condition. Data entered in this section represent individuals, not dyads. Child demographics were collected but only parent outcomes analyzed.
  Participants
    parent: number analyzed (Participants) | 109 | 108 | 105 | 322
    parent: Hispanic or Latino | 9 | 10 | 8 | 27
    parent: Not Hispanic or Latino | 100 | 98 | 97 | 295
    parent: Unknown or Not Reported | 0 | 0 | 0 | 0
    child: number analyzed (Participants) | 109 | 108 | 105 | 322
    child: Hispanic or Latino | 21 | 22 | 10 | 53
    child: Not Hispanic or Latino | 88 | 86 | 95 | 269
    child: Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: At baseline there were 109 parent-child dyads in the web/ mobile-only condition, 108 dyads in the web/ mobile + coach condition, and 105 dyads in the wait list control condition. Data entered in this section represent individuals, not dyads. Child demographics were collected but only parent outcomes analyzed.
  Participants
    parent: number analyzed (Participants) | 109 | 108 | 105 | 322
    parent: American Indian or Alaska Native | 2 | 3 | 1 | 6
    parent: Asian | 3 | 1 | 0 | 4
    parent: Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
    parent: Black or African American | 4 | 2 | 1 | 7
    parent: White | 87 | 86 | 94 | 267
    parent: More than one race | 6 | 10 | 3 | 19
    parent: Unknown or Not Reported | 7 | 5 | 6 | 18
    child: number analyzed (Participants) | 109 | 108 | 105 | 322
    child: American Indian or Alaska Native | 1 | 3 | 1 | 5
    child: Asian | 3 | 0 | 1 | 4
    child: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    child: Black or African American | 4 | 1 | 1 | 6
    child: White | 78 | 78 | 85 | 241
    child: More than one race | 14 | 16 | 12 | 42
    child: Unknown or Not Reported | 9 | 10 | 5 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 218 | 216 | 210 | 644
Family Socioeconomic Status (SES) Risk [Mean (Standard Deviation); unit: score on a scale] — Cumulative risk index (range 0-6) measuring multiple risk factors. The index is based on six dichotomous demographic indicators: the parent does not have a high school diploma or GED, the parent is single, the parent's income is below the poverty threshold (relative to family size), the parent is a recipient of financial assistance (e.g., food stamps), the parent is currently unemployed, or the family's home is overcrowded (i.e., in the bottom one-third of the sample for room-to-occupant ratio). A higher score indicates higher cumulative risk. Population: This variable was only collected from one member of each parent-child dyad (specifically, it was collected from the parent), so the row population is 1/2 of the overall population in which parents and children were combined.
  score on a scale
    number analyzed (Participants) | 109 | 108 | 105 | 322
    (all) | 0.99 (1.17) | 1.20 (1.39) | 0.90 (1.11) | 1.03 (1.23)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Youth Effortful Control Across 12 Months (Parent Report)
Description: Parents reported on their child's effortful attention control via questionnaire using an 8-item subscale of the Early Adolescent Temperament Questionnaire- Revised. Parents were asked to use a 5-pt scale with endpoints of "almost always untrue" and "almost always true" to indicate how well each of 8 statements described their child. Scores ranged from 1-5. High scores indicate greater self-regulation.
Time Frame: baseline; 3 months; 6 months; 1 year
Population: Number of participants differs between baseline and follow-up waves due to attrition (e.g., participants not returning follow-up surveys).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web/ Mobile-only | Web/Mobile + Coach | Wait List Control
Number analyzed (Participants) | 109 | 108 | 105
score on a scale
  Baseline | 3.37 (0.92) | 3.19 (0.91) | 3.34 (0.95)
  3-month follow-up: number analyzed (Participants) | 101 | 98 | 103
  3-month follow-up | 3.39 (0.88) | 3.36 (0.85) | 3.29 (0.95)
  6-month follow-up: number analyzed (Participants) | 102 | 95 | 101
  6-month follow-up | 3.44 (0.84) | 3.36 (0.86) | 3.33 (0.88)
  12-month follow-up: number analyzed (Participants) | 102 | 92 | 99
  12-month follow-up | 3.33 (0.8) | 3.31 (0.92) | 3.21 (0.92)
Statistical Analysis 1: Comparison: Web/ Mobile-only vs Wait List Control; Test type: Superiority; p = .549, t-test, 2 sided; Mean Difference (Final Values) = 0.07 — Mean difference in slope with the wait-list control as the reference group
Statistical Analysis 2: Comparison: Web/Mobile + Coach vs Wait List Control; Test type: Superiority; p = .854, t-test, 2 sided; Mean Difference (Final Values) = -0.02 — Mean difference in slope with the wait-list control as the reference group
Statistical Analysis 3: Comparison: Web/ Mobile-only vs Web/Mobile + Coach; Test type: Superiority; p = .469, t-test, 2 sided; Mean Difference (Final Values) = -0.09 — Mean difference in slope with the web/mobile only as the reference group

2. Primary Outcome: Change From Baseline in Sense of Parenting Importance Across 12 Months (Parent Report)
Description: Using a measure developed for the purposes of this study, parents were provided with a list of 14 parenting skills that closely corresponded to skills that were supported in the FCU Online parenting curriculum, shich as "providing praise and encouragement for good behavior" and "setting clear rules and expectations for behavior." For each parenting skill, parents were asked to indicate the importance of this skill during the middle school years using a 5-point scale with endpoints of "not at all important" and "very important." Scores ranged from 1-5. Higher scores indicate higher endorsement of the importance of parenting skills.
Time Frame: baseline; 3 months; 6 months; 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web/ Mobile-only | Web/Mobile + Coach | Wait List Control
Number analyzed (Participants) | 109 | 108 | 105
score on a scale
  baseline | 4.51 (0.31) | 4.55 (0.24) | 4.49 (0.30)
  3-month follow-up: number analyzed (Participants) | 101 | 98 | 103
  3-month follow-up | 4.48 (0.35) | 4.59 (0.27) | 4.47 (0.31)
  6-month follow-up: number analyzed (Participants) | 102 | 95 | 101
  6-month follow-up | 4.51 (0.34) | 4.56 (0.29) | 4.47 (0.30)
  12-month follow-up: number analyzed (Participants) | 102 | 92 | 99
  12-month follow-up | 4.48 (0.34) | 4.55 (0.29) | 4.47 (0.32)
Statistical Analysis 1: Comparison: Web/ Mobile-only vs Wait List Control; Test type: Superiority; p = .535, t-test, 2 sided; Mean Difference (Final Values) = 0.03 — Mean difference in slope with the wait-list control as the reference group
Statistical Analysis 2: Comparison: Web/Mobile + Coach vs Wait List Control; Test type: Superiority; p = .081, t-test, 2 sided; Mean Difference (Final Values) = 0.08 — Mean difference in slope with the wait-list control as the reference group
Statistical Analysis 3: Comparison: Web/ Mobile-only vs Web/Mobile + Coach; Test type: Superiority; p = .295, t-test, 2 sided; Mean Difference (Final Values) = .05 — Mean difference in slope with the web/mobile only as the reference group

3. Primary Outcome: Change From Baseline in Sense of Parenting Confidence Across 12 Months (Parent Report)
Description: Using a measure developed for the purposes of this study, parents were provided with a list of 14 parenting skills that closely corresponded to skills that were supported in the FCU Online parenting curriculum, shich as "providing praise and encouragement for good behavior" and "setting clear rules and expectations for behavior." For each parenting skill, parents were asked to indicate their level of confidence in using each skill with their child using a 5-point scale with endpoints of "not at all confident" and "very confident." Scores ranged from 1 to 5. Higher scores indicate greater confidence in using parenting skills.
Time Frame: baseline; 3 months; 6 months; 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web/ Mobile-only | Web/Mobile + Coach | Wait List Control
Number analyzed (Participants) | 109 | 108 | 105
score on a scale
  baseline | 4.16 (0.64) | 4.11 (0.51) | 4.13 (0.54)
  3-month follow-up: number analyzed (Participants) | 101 | 98 | 103
  3-month follow-up | 4.23 (0.56) | 4.17 (0.55) | 4.08 (0.62)
  6-month follow-up: number analyzed (Participants) | 102 | 95 | 101
  6-month follow-up | 4.21 (0.54) | 4.20 (0.53) | 4.10 (0.52)
  12-month follow-up: number analyzed (Participants) | 102 | 92 | 99
  12-month follow-up | 4.15 (0.58) | 4.19 (0.54) | 4.03 (0.55)
Statistical Analysis 1: Comparison: Web/ Mobile-only vs Wait List Control; Test type: Superiority; p = .149, t-test, 2 sided; Mean Difference (Final Values) = 0.11 — Mean difference in slope with the wait-list control as the reference group
Statistical Analysis 2: Comparison: Web/Mobile + Coach vs Wait List Control; Test type: Superiority; p = .207, t-test, 2 sided; Mean Difference (Final Values) = 0.10 — Mean difference in slope with the wait-list control as the reference group
Statistical Analysis 3: Comparison: Web/ Mobile-only vs Web/Mobile + Coach; Test type: Superiority; p = .871, t-test, 2 sided; Mean Difference (Final Values) = -0.01 — Mean difference in slope with the web/mobile only as the reference group

4. Primary Outcome: Change From Baseline in Parenting Self-Efficacy Across 12 Months (Parent Report)
Description: Parenting self-efficacy was assessed with 8 self-report items adapted from the Parenting Task Checklist. Using a 5-pt scale with endpoints of "not confident at all" and "very confident," parents were asked to indicated their level of confidence in handling 8 negative child behaviors such as "your child arguing with you about rules" and "your child's mood swings." Scores ranged from 0 to 4. Higher scores indicate greater parenting confidence/ self-efficacy.
Time Frame: baseline; 3 months; 6 months; 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web/ Mobile-only | Web/Mobile + Coach | Wait List Control
Number analyzed (Participants) | 109 | 108 | 105
score on a scale
  baseline | 2.85 (0.79) | 2.66 (0.74) | 2.75 (0.78)
  3-month follow-up: number analyzed (Participants) | 100 | 98 | 103
  3-month follow-up | 2.80 (0.76) | 2.85 (0.70) | 2.75 (0.75)
  6-month follow-up: number analyzed (Participants) | 102 | 95 | 101
  6-month follow-up | 2.90 (0.7) | 2.86 (0.71) | 2.78 (0.75)
  12-month follow-up: number analyzed (Participants) | 101 | 92 | 99
  12-month follow-up | 2.85 (0.73) | 2.91 (0.65) | 2.81 (0.80)
Statistical Analysis 1: Comparison: Web/ Mobile-only vs Wait List Control; Test type: Superiority; p = .547, t-test, 2 sided; Mean Difference (Final Values) = 0.06 — Mean difference in slope with the wait-list control as the reference group
Statistical Analysis 2: Comparison: Web/Mobile + Coach vs Wait List Control; Test type: Superiority; p = .575, t-test, 2 sided; Mean Difference (Final Values) = 0.06 — Mean difference in slope with the wait-list control as the reference group
Statistical Analysis 3: Comparison: Web/ Mobile-only vs Web/Mobile + Coach; Test type: Superiority; p = .964, t-test, 2 sided; Mean Difference (Final Values) = 0.00 — Mean difference in slope with the web/mobile only as the reference group

5. Primary Outcome: Change From Baseline in Youth Conduct Problems Across 12 Months (Parent Report)
Description: Parents reported on their child's problem behavior using the Strengths and Difficulties Questionnaire (SDQ), a 25-item brief behavioral screening questionnaire that consists of 5 subscales with 5 questions each. The 5 subscales are conduct problems, emotional problems, hyperactivity, peer problems, and prosocial behavior. Parents were asked to indicate the extent to which statements were true of their child's behavior in the past month using a 3-pt scale (not true, somewhat true, and certainly true). The conduct problems subscale included items such as "often loses temper" and "often fights with other youth or bullies them." Scores ranged from 0 to 10. High scores indicate greater conduct problems.
Time Frame: baseline; 3 months; 6 months; 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web/ Mobile-only | Web/Mobile + Coach | Wait List Control
Number analyzed (Participants) | 109 | 108 | 105
score on a scale
  Baseline | 1.37 (1.81) | 1.44 (1.65) | 1.05 (1.38)
  3-month follow-up: number analyzed (Participants) | 101 | 98 | 103
  3-month follow-up | 1.32 (1.63) | 1.30 (1.55) | 1.24 (1.54)
  6-month follow-up: number analyzed (Participants) | 102 | 95 | 101
  6-month follow-up | 1.17 (1.57) | 1.12 (1.54) | 1.00 (1.44)
  12-month follow-up: number analyzed (Participants) | 102 | 92 | 99
  12-month follow-up | 1.19 (1.40) | 1.21 (1.60) | 1.08 (1.45)
Statistical Analysis 1: Comparison: Web/ Mobile-only vs Wait List Control; Test type: Superiority; p = .236, t-test, 2 sided; Mean Difference (Final Values) = 0.04 — Mean difference in slope with the wait-list control as the reference group
Statistical Analysis 2: Comparison: Web/Mobile + Coach vs Wait List Control; Test type: Superiority; p = .142, t-test, 2 sided; Mean Difference (Final Values) = 0.05 — Mean difference in slope with the wait-list control as the reference group
Statistical Analysis 3: Comparison: Web/ Mobile-only vs Web/Mobile + Coach; Test type: Superiority; p = .810, t-test, 2 sided; Mean Difference (Final Values) = 0.01 — Mean difference in slope with the web/mobile only as the reference group

6. Primary Outcome: Change From Baseline in Youth Hyperactivity Across 12 Months (Parent Report)
Description: Parents reported on their child's problem behavior using the Strengths and Difficulties Questionnaire (SDQ), a 25-item brief behavioral screening questionnaire that consists of 5 subscales with 5 questions each. The 5 subscales are conduct problems, emotional problems, hyperactivity, peer problems, and prosocial behavior. Parents were asked to indicate the extent to which statements were true of their child's behavior in the past month using a 3-pt scale (not true, somewhat true, and certainly true). The hyperactivity subscale included items such as "restless, overactive, cannon sit still for long" and "easily distracted, concentration wanders." Scores ranged from 0 to 10. High scores indicate greater hyperactivity.
Time Frame: baseline; 3 months; 6 months; 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web/ Mobile-only | Web/Mobile + Coach | Wait List Control
Number analyzed (Participants) | 109 | 108 | 105
score on a scale
  baseline | 3.72 (2.46) | 4.19 (2.87) | 3.45 (2.69)
  3-month follow-up: number analyzed (Participants) | 101 | 98 | 103
  3-month follow-up | 3.20 (2.02) | 3.47 (2.39) | 3.31 (3.43)
  6-month follow-up: number analyzed (Participants) | 102 | 95 | 101
  6-month follow-up | 3.11 (2.39) | 3.45 (2.37) | 3.24 (2.32)
  12-month follow-up: number analyzed (Participants) | 102 | 92 | 99
  12-month follow-up | 3.21 (2.10) | 3.41 (2.47) | 3.46 (2.56)
Statistical Analysis 1: Comparison: Web/ Mobile-only vs Wait List Control; Test type: Superiority; p = .599, t-test, 2 sided; Mean Difference (Final Values) = -0.17 — Mean difference in slope with the wait-list control as the reference group
Statistical Analysis 2: Comparison: Web/Mobile + Coach vs Wait List Control; Test type: Superiority; p = .523, t-test, 2 sided; Mean Difference (Final Values) = 0.22 — Mean difference in slope with the wait-list control as the reference group
Statistical Analysis 3: Comparison: Web/ Mobile-only vs Web/Mobile + Coach; Test type: Superiority; p = .252, t-test, 2 sided; Mean Difference (Final Values) = 0.36 — Mean difference in slope with the web/mobile only as the reference group

7. Primary Outcome: Change From Baseline in Youth Emotional Problems Across 12 Months (Parent Report)
Description: Parents reported on their child's problem behavior using the Strengths and Difficulties Questionnaire (SDQ), a 25-item brief behavioral screening questionnaire that consists of 5 subscales with 5 questions each. The 5 subscales are conduct problems, emotional problems, hyperactivity, peer problems, and prosocial behavior. Parents were asked to indicate the extent to which statements were true of their child's behavior in the past month using a 3-pt scale (not true, somewhat true, and certainly true). The emotional problems subscale included items such as "many worries or often seemed worried" and "often unhappy, depressed, or tearful." Scores ranged from 0 to 10. High scores indicate greater emotional problems.
Time Frame: baseline; 3 months; 6 months; 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web/ Mobile-only | Web/Mobile + Coach | Wait List Control
Number analyzed (Participants) | 109 | 108 | 105
score on a scale
  Baseline | 2.56 (2.28) | 2.78 (2.12) | 2.34 (2.27)
  3-month follow-up: number analyzed (Participants) | 101 | 98 | 103
  3-month follow-up | 2.36 (2.23) | 2.20 (1.97) | 2.56 (2.42)
  6-month follow-up: number analyzed (Participants) | 102 | 95 | 101
  6-month follow-up | 2.45 (2.37) | 2.31 (2.04) | 2.47 (2.30)
  12-month follow-up: number analyzed (Participants) | 102 | 92 | 99
  12-month follow-up | 2.64 (2.43) | 2.09 (1.96) | 2.60 (2.37)
Statistical Analysis 1: Comparison: Web/ Mobile-only vs Wait List Control; Test type: Superiority; p = .867, t-test, 2 sided; Mean Difference (Final Values) = 0.06 — Mean difference in slope with the wait-list control as the reference group
Statistical Analysis 2: Comparison: Web/Mobile + Coach vs Wait List Control; Test type: Superiority; p = .127, t-test, 2 sided; Mean Difference (Final Values) = -0.47 — Mean difference in slope with the wait-list control as the reference group
Statistical Analysis 3: Comparison: Web/ Mobile-only vs Web/Mobile + Coach; Test type: Superiority; p = .101, t-test, 2 sided; Mean Difference (Final Values) = -0.51; Mean difference in slope with the web/mobile only as the reference group

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events over the study period (until their 12-month post-test was completed).
Arm/Group | Web/ Mobile-only | Web/Mobile + Coach | Wait List Control
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/108 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/108 | 0/105
Other Adverse Events (participants affected / at risk) | 0/109 | 0/108 | 0/105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT03060291/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/91/NCT03060291/SAP_001.pdf
  • Informed Consent Form (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/91/NCT03060291/ICF_002.pdf